CLINICAL TRIAL: NCT05403047
Title: Efficacy of Tenofovir Disoproxil on Mother-to-child Transmission of HBV in Tokombéré, Cameroon in Pregnant Women Infected With Hepatitis B Virus (HBeAg Positive or With a High Viral Load) and Whose Newborns Had Been Vaccinated at Birth
Brief Title: Efficacy of Tenofovir Disoproxil on Mother-to-child Transmission of HBV in Tokombéré, Cameroon in Pregnant Women
Acronym: TOPCHIB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Principal Investigator, dourwe maaga, head of the ANRS 12417 project, ANRS, Emerging Infectious Diseases
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 12417 TOPCHIB
Record Dates: First submitted 2022-05-23; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis B Virus - Chronic Active
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- pregnant woman - tenofovir (Other): Participants will be started on tenofovir disoproxil fumarate (TDF) 245 mg one tablet per day from week 28 of pregnancy until 6 weeks postpartum.
  Interventions: Drug: Fumarate, Tenofovir Disoproxil

INTERVENTIONS:
Drug: Fumarate, Tenofovir Disoproxil — all participants receive the intervention
  Other Names: TDF

SUMMARY:
IIn this study, pregnant women with HBeAg-positive viral hepatitis b or high viral load will receive Tenofovir disoproxil fumarate from the 28th week of amenorrhoea until 6 weeks after delivery. Their newborns will receive the hepatitis B vaccine, starting with one dose at birth and followed by three booster doses, according to the Expanded Programme on Immunisation. The investigators hypothesise that a short course of TDF could greatly reduce the risk of HBV MTCT in pregnant women at high risk of MTCT (HBeAg positive or with high viral load).

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label, descriptive, phase IV clinical trial in HBsAg and HBeAg positive pregnant women. Eligible pregnant women will receive 245 mg of tenofovir disoproxil fumarate once daily from 28 weeks of pregnancy until 6 weeks after delivery. Newborns will receive the hepatitis B vaccine, starting with one dose at birth, followed by three booster doses, in accordance with the expanded programme of vaccination.

The study aims to show that the addition of maternal antiviral treatment to vaccination at birth followed by three booster doses can be favourably considered in the context where vaccination alone is not sufficient to prevent transmission of the hepatitis B virus from mother to child. A total of 150 pregnant women will be included in the Tokombéré district.

ELIGIBILITY:
Inclusion criteria:

* Pregnant women with a term of less than 24 weeks of amenorrhea;
* HBsAg positive ;
* HBeAg positive or HBeAg negative with a high viral load ( > 200 000 UI/ml) ;
* 16 years old or more on the inclusion day ;
* Signature of free and informed consent (for pregnant women aged 16 to 21, the participant's consent as well as the authorization of a parent/adult husband/ legal tutor will be collected) which also includes consent for the children

Exclusion criteria :

* HIV co-infection;
* Women treated for HBV;
* Creatinine clearance <30 ml / min;
* Suspicion of poor monitoring of children's vaccination schedule for HBV (vaccination at birth + boosters);
* Disease or treatment contraindicating the taking of TDF.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant woman
Enrollment: 150 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of children with HBsAg positive at 9-12 months of life (W36 - W48) in the study population, | measured between 36 and 48 weeks of life of the child of the mothers included in the study
  Proportion of HBsAg-positive children between 9 and 12 months of age in the study population, assessed by an automated test (mini VIDAS)

CONTACTS AND LOCATIONS:
Overall Officials: Pr Yazdan YAZDANPANAH, Study Director — ANRS, Emerging Infectious Diseases

IPD SHARING:
Plan to Share IPD: Undecided